CLINICAL TRIAL: NCT00638820
Title: Reduced Intensity Allogeneic Transplantation For Severe Osteopetrosis Incorporating A Second Cd34 Selected Graft
Brief Title: Reduced Intensity AlloTransplant For Osteopetrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Excess toxicity
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Paul Orchard, M.D., University of Minnesota
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0704M06581; MT2007-06 (Other: Masonic Cancer Center, University of Minnesota)
Record Dates: First submitted 2008-03-11; First posted 2008-03-19 (Estimated); Results first posted 2010-02-03 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Osteopetrosis
Keywords: osteopetrosis
MeSH Terms: conditions — Osteopetrosis | interventions — Cord Blood Stem Cell Transplantation; Bone Marrow Transplantation; Alemtuzumab; Busulfan; Clofarabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intent-To-Treat (Experimental): Patients enrolled and received study treatment.
  Interventions: Procedure: Stem Cell or Umbilical Cord Blood Transplantation; Drug: Campath, Busulfan, Clofarabine; Procedure: Total Lymphoid Irradiation

INTERVENTIONS:
Procedure: Stem Cell or Umbilical Cord Blood Transplantation — Stem Cell (unrelated or matched related donor grafts (both peripheral blood and marrow) infusion on Day 0 and 42; Umbilical Cord Blood on Day 0 and 42
  Other Names: Bone Marrow Transplant
Drug: Campath, Busulfan, Clofarabine — * 12 Campath-1H 0.3 mg/kg intravenously (IV) over 2 hours
  * 11 Campath-1H 0.3 mg/kg intravenously over 2 hours
  * 10 Campath-1H 0.3 mg/kg intravenously over 2 hours
  * 9 Busulfan <12 kg: 2.2 mg/kg/dose IV every 12 hours >12 kg: 1.6 mg/kg/dose IV every 12 hours
  * 8 Busulfan <12 kg: 2.2 mg/kg/dose IV every 12 hours >12 kg: 1.6 mg/kg/dose IV every 12 hours
  * 7 "Rest"
  * 6 Clofarabine 40 mg/m2 intravenously over 2 hours
  * 5 Clofarabine 40 mg/m2 intravenously over 2 hours
  * 4 Clofarabine 40 mg/m2 intravenously over 2 hours
  * 3 Clofarabine 40 mg/m2 intravenously over 2 hours
  * 2 Clofarabine 40 mg/m2 intravenously over 2 hours
  Other Names: Busulfex, Clolar,Alemtuzumab
Procedure: Total Lymphoid Irradiation — Dose 500 cGy via anteroposterior (AP) and posteroanterior (PA) fields (250 cGy AP and 250 cGy PA).
  Other Names: Therapuetic radation, radiation therapy

SUMMARY:
We believe that hematopoietic stem cell transplantation (HSCT) will help subjects with Osteopetrosis generate functioning osteoclasts, and by so doing assist in the resolution of the abnormal bone architecture, and the anemia and bone marrow failure that is also characteristic of this disease. However, we have found in past studies that approximately 30% of Osteopetrosis patients do not engraft. Therefore, in this study, we plan to use a different combination of pre-transplant drugs to try to make transplants safer for this disease, as well as to provide a second infusion of stem cells in patients with matched related or unrelated donors. The purpose of this research is to find a safer and more effective means of performing stem cell transplantation in patients with Osteopetrosis, using chemotherapy and radiation designed to bring about engraftment and lessen transplant mortality.

DETAILED DESCRIPTION:
This transplant protocol will test the following: 1) the ability to achieve engraftment with the reduced intensity protocol, 2) the mortality associated with transplant by day 100, 3) patient outcomes, based on differential imaging and biologic evaluations prior to transplantation and at designated points after transplantation (day 100, 6 months, 1, 2 and 5 years). Additional biologic studies will include microarray analysis, Campath levels just prior to the administration of the graft, and establishment of mesenchymal stem cell lines. In older patients, studies to evaluation osteoclast differentiation and function will also be offered.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for transplantation under this protocol will be <45 years of age, and will be diagnosed with severe osteopetrosis. This will be defined as having the following manifestations of the disease.
* Bones that are uniformly markedly dense based on skeletal survey
* No history that would suggest autosomal dominant inheritance
* Evidence of hematologic changes that are attributed to the underlying disease, including the need for ongoing transfusions, OR
* the presence of progressive anemia or thrombocytopenia, OR a white blood cell differential with a predominance of immature forms and evidence of extramedullary hematopoiesis, OR
* persistence of serious infectious complications that are thought to be due to the abnormal architecture of the bone that are resistant to surgical and medical interventions.

Exclusion Criteria:

* Patients >45 years of age
* Evidence of hepatic failure
* pulmonary dysfunction sufficient to substantially increase the risk of transplant
* Renal dysfunction with glomerular filtration rate (GFR) <30% of predicted.
* Cardiac compromise sufficient to substantially increase the risk of transplantation
* Severe, stable neurologic impairment.
* Human immunodeficiency virus (HIV) positivity.
* Pregnant or lactating females

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of MInnesota, Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated early due to stopping rules. The first 3 patients enrolled died by Day 100 of study.
Groups:
- Patients With Osteopetrosis Who Received Transplant: All patients enrolled with osteopetrosis and received transplant.
Period: Overall Study
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Donor Cell Engraftment
Description: Number of patients with persistent presence of donor-derived cells at Day 100
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Number analyzed (Participants) | 3
Participants | 2

2. Secondary Outcome: Number of Patients With Transplant Related Death
Description: Number of participants died during study by Day 100 and reason for death was related to transplant.
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Number of Patients With Transplant Related Toxicity
Description: Number of patients experiencing adverse effects due to transplant categorized by body system using Common Terminology Criteria for Adverse Events coding from the National Cancer Institute, Version 3.0.
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Number analyzed (Participants) | 3
Participants
  Neurologic | 1
  Renal | 1
  Pulmonary | 3
  Peri-Transplant Mortality (Death by Day 100) | 3
  Vascular | 1

4. Secondary Outcome: Differential Imaging and Biologic Evaluations
Description: These outcome measures were not assessed due to early study termination.
Time Frame: Day 100, 6 months, 1, 2 and 5 years
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 through Day 100 of the study.
Arm/Group | Patients With Osteopetrosis Who Received Transplant
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Osteopetrosis Who Received Transplant (N=3)
Death, peri-transplant (General disorders) | 3 (3) — Death was related to receiving transplant.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Osteopetrosis Who Received Transplant (N=3)
Neurologic (Nervous system disorders) | 1 (1)
Renal (Renal and urinary disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vascular (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only 3 participants were treated in this study; all died by Day 100. Data for both treatment arms were combined due to low number. (Arm 1 utilized mobilized peripheral blood or marrow (related or unrelated). Arm 2 received cord blood transplants).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes